CLINICAL TRIAL: NCT06644924
Title: A Phase II, Randomized, Double-blind, Single-dose, Placebo-controlled, 3-Period, 3-Treatment, Crossover, Multicenter Study to Compare the Bronchodilatory Effect and Safety of PT007 to Placebo MDI and Open-Label Ventolin® Evohaler in Adult Participants With Asthma
Brief Title: A Study Evaluating the Effect of Inhaled PT007(AS MDI) Versus Placebo MDI and Ventolin Evohaler on Lung Function in Adult Participants With Asthma
Acronym: MITCHELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6935C00002
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Asthma, Bronchial; Bronchial Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Anti-Asthmatic Agents; Respiratory System Agents
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AS MDI and placebo MDI will be blinded to all participants, study site staff, endpoint assessors, and sponsor personnel. Placebo MDI is designed to mimic the appearance, smell, and taste of AS MDI. No double-dummy will be used. Packaging and labelling of AS MDI and placebo MDI will be designed to ensure blinding.
  The IRT will provide to the investigator(s) or pharmacist(s) the kit identification number to be allocated to the participant at the dispensing visits. Routines for this will be described in the IRT user manual that will be provided to each study site.
  Randomized Ventolin Evohaler is open label. However, to reduce bias, dosing will be performed under the supervision of study staff, and spirometry assessments will be performed by different study personnel who will only enter the room after dosing is completed; thus, the study personnel conducting the spirometry assessments will be blinded to the identity of the study intervention."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Treatment Sequence 1 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment A (Ventolin Evohaler) , Treatment B (Placebo MDI), and Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI
- Treatment Sequence 2 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), Treatment A (Ventolin Evohaler) and Treatment B (Placebo MDI).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI
- Treatment Sequence 3 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment B (Placebo MDI), Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), Treatment A (Ventolin Evohaler).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI
- Treatment Sequence 4 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), Treatment B (Placebo MDI), Treatment A (Ventolin Evohaler).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI
- Treatment Sequence 5 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment B (Placebo MDI), Treatment A (Ventolin Evohaler), and Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI
- Treatment Sequence 6 (Experimental): Participants will be randomized to 1 of the 6 different treatment sequences. Each treatment sequence consist of Treatment A (Ventolin Evohaler), Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007) and Treatment B (Placebo MDI).
  Interventions: Combination Product: Intervention: AS MDI; Combination Product: Intervention: Ventolin Evohaler; Combination Product: Intervention: Placebo matching AS MDI

INTERVENTIONS:
Combination Product: Intervention: AS MDI — Drug Treatment: (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007) Randomized participants will receive a single-dose (2 inhalations)
  Other Names: Albuterol Sulfate metered dose inhaler [AS MDI] - PT007)
Combination Product: Intervention: Ventolin Evohaler — Drug: Treatment (Ventolin Evohaler) Randomized participants will receive a single-dose (2 inhalations)
Combination Product: Intervention: Placebo matching AS MDI — Drug: Treatment (Placebo MDI) Randomized participants will receive a single-dose (2 inhalations to match AS MDI)

SUMMARY:
Phase II study, to investigate the therapeutic efficacy and safety of inhaled PT007 (referred to as AS MDI) compared with placebo MDI and open-label Ventolin Evohaler in male and female participants aged 18 to 65 years (inclusive) with asthma.

This study consists of a screening/run-in period, a treatment period, and a follow-up phone call.

DETAILED DESCRIPTION:
This is a randomized, double-blind, single-dose, placebo-controlled, 3-period, 3-treatment, crossover, multicenter study to assess the bronchodilatory effect and safety of AS MDI (180 μg) compared with placebo MDI and open-label Ventolin Evohaler (200 μg) in adult participants (aged 18 to 65 years, inclusive) with asthma (pre-bronchodilator FEV1 of ≥ 40% of the predicted normal value) and demonstrated FEV1 reversibility to Ventolin hydrofluoroalkane (HFA) (improvement in FEV1 at 30 minutes post-Ventolin HFA dosing of ≥ 12% and ≥ 200 mL).

The study duration will be a minimum of 15 days and up to a maximum of 52 days.

Including:

screening/run-in period: 3 to 28 days treatment period: 9 to 17 days follow-up phone call: 3 to 7 days after the final dose of study intervention

Eligible participants will be randomized to 1 of 6 predefined treatment sequences in a 1:1:1:1:1:1 ratio. Each sequence will contain AS MDI, placebo MDI, and Ventolin Evohaler in a randomized order.

Eligible participants will receive a single dose of randomized study intervention at each of 3 treatment visits (Visits 2, 3, and 4), with a 3- to 7-day washout period between treatment visits.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be aged 18 to 65 years (inclusive), at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants should have a documented history of physician-diagnosed asthma ≥ 6 months prior to Visit 1.
3. Must be receiving one of the following required inhaled asthma therapies listed below for at least the last 30 days:

   1. Only SABA, which is used as needed for rescue.
   2. Low to medium doses of ICS (alone or in combination with LABA), used regularly as maintenance asthma therapy.
4. Pre-BD FEV1 of ≥ 40% of the PN value at Visit 1, after withholding SABA for ≥ 6 hours (and Visit 1a and/or Visit 1b, if applicable).
5. Confirmed FEV1 reversibility to 4 actuations of Ventolin HFA, defined as a post-Ventolin HFA increase in FEV1 at 30 minutes of ≥ 12% and ≥ 200 mL at either Visit 1, Visit 1a, or Visit 1b; only 2 reversibility testing attempts are allowed.
6. Demonstrate acceptable spirometry performance (ie, meet ATS/ERS acceptability/repeatability criteria).
7. Willing and, in the opinion of the investigator, able to adjust current asthma therapy, as required by the protocol.
8. Demonstrate acceptable MDI administration technique. Note: Use of a spacer device during the screening and randomized treatment periods is not permitted.

   Weight
9. Body mass index < 40 kg/m2. Sex and Contraceptive/Barrier Requirements
10. Contraceptive use by females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
11. Female participants: A participant of childbearing potential, must have a negative urine pregnancy test at Visit 1 (to be read locally).

    Participants not of childbearing potential are defined as those who are physiologically incapable of becoming pregnant, including any participant who is 2 years postmenopausal, or surgically sterile (defined as having a bilateral oophorectomy, hysterectomy, tubal ligation, or other permanent birth control measures).

    Participants aged ≥ 50 years will be considered postmenopausal if they have been amenorrheic for 12 consecutive months or more following cessation of all exogenous hormonal treatment.

    Participants aged < 50 years will be considered postmenopausal if they have been amenorrheic for 12 consecutive months or more following cessation of exogenous hormonal treatment and in the absence of any alternative medical cause, as judged by the investigator.
12. Participants of childbearing potential must use a highly effective form of contraception from signing of the ICF to 14 days after the last study intervention. Highly effective birth control methods are listed below:

    Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).

    Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation):
    * Oral
    * Intravaginal (eg, NuvaRing®)
    * Transdermal (eg, Evra Patch™, Xulane™)

    Progestogen-only hormonal contraception associated with inhibition of ovulation:
    * Oral
    * Injectable (eg, Depo-Provera™)
    * Implantable (eg, Implanon®) Intrauterine device or intrauterine hormone-releasing system Bilateral tubal occlusion Male partner sterilization/vasectomy with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis, or medical history interview provided by her or her partner.

    Note: Periodic abstinence (calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), declaration of abstinence for the duration of exposure to study intervention, spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

    Informed Consent
13. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

    Other Inclusion Criteria
14. Compliance: must be willing to remain at the study site as required per protocol to complete all visit assessments.

Exclusion Criteria:

5.2 Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions and History

1. Any evidence of chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or that could affect the efficacy or safety analysis.
2. Life-threatening asthma defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s) within the last 5 years.
3. Upper respiratory infection not resolved within 7 days of Visit 1 and throughout the screening period.
4. Hospitalizations for asthma exacerbation within the last 3 months prior to Visit 1.
5. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (eg, congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia, participants with known QTcF ≥ 480 ms, coronary heart disease), hepatic, renal, hematological, neuropsychological, endocrine (eg, uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), or gastrointestinal (eg, poorly controlled peptic ulcer, gastroesophageal reflux disease). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through study participation, or that could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
6. Cancer not in complete remission for at least 5 years prior to Visit 1. Note: Participants with squamous cell carcinoma of the skin or basal cell carcinoma of the skin or cervical carcinoma in situ are eligible, if in the opinion of the investigator, the condition has been adequately worked up and clinically controlled, and the participant's participation in the study would not represent a safety concern.
7. Hospitalized for psychiatric disorder or attempted suicide within one year prior to Visit 1.
8. History of psychiatric disease, intellectual deficiency, poor motivation, or other conditions limiting informed consent validity.
9. Received a live attenuated vaccination within 7 days of Visit 1. Prior/Concomitant Therapy
10. Oral/systemic corticosteroid use (any dose) within 6 weeks of Visit 1.
11. Chronic use of oral corticosteroids (≥ 3 weeks use in the 3 months prior to Visit 1).
12. Received any marketed (eg, omalizumab, mepolizumab, reslizumab) or investigational biologic within 3 months or 5 half-lives, whichever is longer, or any other medication specifically prohibited by the protocol within the indicated exclusionary time periods.
13. Received tiotropium within 2 weeks of Visit 1.
14. Received treatment for lower respiratory infection or asthma exacerbation within 6 weeks of Visit 1.
15. Unable to abstain from protocol-defined prohibited medications during screening and the study.
16. Using any herbal products by inhalation or nebulizer within 2 weeks of Visit 1 and does not agree to stop during the study duration.

    Prior/Concurrent Clinical Study Experience
17. Treatment with investigational study intervention (or device) in another clinical study within the last 30 days or 5 half-lives, whichever is longer, prior to Visit 1.
18. Hypersensitivity to β2-agonists or any component of the investigational MDI or any component of Ventolin Evohaler or HFA (or Pulmicort Flexhaler, if applicable).

    Other Exclusions
19. Significant abuse of alcohol or drugs in the opinion of the investigator.
20. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months (including all forms of tobacco, e-cigarettes [vaping], and marijuana).
21. Study investigators, sub-investigators, coordinators, and their employees or immediate family members, or employees of the sponsor.
22. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
23. For female participants only: currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FEV1 AUC 0-6 hours | 0 to 6 hours (Spirometry will be obtained 60 and 30 minutes pre-dose and 5, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes post-dose)
  Change from baseline FEV1 measured at each time point. Baseline FEV1 is the period specific mean of the available pre-dose values. Area Under the Curve (AUC) is calculated for the available time points using the trapezoidal rule.

SECONDARY OUTCOMES:
Change from baseline in FEV1 AUC 0 - 4 hours | 0 to 4 hours (Spirometry will be obtained at 5, 15, 30, 45, 60, 120, 180, and 240 minutes post-dose)
  Change from baseline FEV1 measured at each time point. Baseline FEV1 is the period specific mean of the available pre-dose values. Area Under the Curve (AUC) is calculated for the available time points using the trapezoidal rule.
Peak Change From Baseline in FEV1 | Over 6 hours post dose
  Peak change from baseline in FEV1 is the maximum change from baseline FEV1 that is measured over the timeframe. Baseline FEV1 is the period specific mean of the available pre-dose values.

OTHER OUTCOMES:
Adverse events (AE)/serious adverse events (SAE) | From randomization throughout the treatment period and including the follow-up period (telephone contact).
  Safety data collected on treatment and on study.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Research Site, Encinitas, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Stockton, California
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, White Marsh, Maryland
  - Research Site, Columbia, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, Victoria, Texas
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Phrma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/